CLINICAL TRIAL: NCT03864978
Title: Safety and Efficacy of Rifaximin Delayed Release 400 mg Tablets in Patients With Moderate-to-severe Papulopustular Rosacea and Positive Lactulose Breath Test. A Multicenter Double-blind, Placebo-controlled Randomized Clinical Trial
Brief Title: Safety and Efficacy of Rifaximin in Patients With Papulopustular Rosacea and Positive Lactulose Breath Test
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REROS/001/17; 2017-003722-33 (EudraCT Number)
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rifaximin-EIR 800 mg BID for 10 days (Experimental): 2 x rifaximin delayed release 400 mg tablet twice a day (total daily dose of rifaximin: 1600 mg) for 10 days and 2 x placebo tablets twice a day for the following 20 days
  Interventions: Drug: Rifaximin delayed release 400 mg tablet; Drug: Placebo
- Rifaximin-EIR 400 mg BID for 30 days (Experimental): 1 x rifaximin delayed release 400 mg tablet + 1 x placebo tablet twice a day (total daily dose of rifaximin: 800 mg) for 30 days
  Interventions: Drug: Rifaximin delayed release 400 mg tablet; Drug: Placebo
- Rifaximin-EIR 400 mg BID for 10 days (Experimental): 1 x rifaximin delayed release 400 mg tablet + 1 x placebo tablet twice a day (total daily dose of rifaximin: 800 mg) for 10 days and 2 x placebo tablets twice a day for the following 20 days
  Interventions: Drug: Rifaximin delayed release 400 mg tablet; Drug: Placebo
- Two placebo tablets BID for 30 days (Placebo Comparator): 2 x placebo tablets twice a day for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin delayed release 400 mg tablet — Rifaximin delayed release
  Arms: Rifaximin-EIR 400 mg BID for 10 days; Rifaximin-EIR 400 mg BID for 30 days; Rifaximin-EIR 800 mg BID for 10 days
Drug: Placebo — Placebo

SUMMARY:
Preliminary evidence suggests that treatment with rifaximin may be beneficial in patients with papulopustular rosacea.

The present clinical trial is aimed to investigate the safety and efficacy of oral rifaximin delayed release versus placebo in adults with moderate-to-severe papulopustular rosacea (a.k.a. subtype II) and positive lactulose H2/CH4 breath test.

ELIGIBILITY:
Key inclusion Criteria:

1. Men and women aged 18 to 70 years at screening.
2. Female participants are eligible if they are either of non-childbearing potential or of childbearing potential with a negative pregnancy test result at screening and randomization and agreeing to use a highly effective method of contraception until 72 hours after taking the last study treatment dose.
3. Moderate-to-severe papulopustular rosacea (a.k.a. subtype II, RII) at screening and confirmed at randomization. Moderate-to-severe rosacea is defined as the presence of 11 or more facial papules or pustules with or without plaques.
4. Positivity of lactulose H2/CH4 breath test (L-BT) within the last 2-weeks before randomization.
5. Patients accepting to provide and legally capable of providing free and informed consent to all procedures included in the protocol (including facial skin photography).

Key exclusion Criteria:

1. Granulomatous rosacea or rosacea fulminans.
2. Erythematoteleangectatic, phymatous or ocular rosacea only. Patients with these subtypes associated with papulopustular rosacea can be enrolled.
3. Circulating anti-helicobacter pylori IgM and/or IgG at screening (V1).
4. Positivity at the faecal Clostridium Difficile toxin assay at screening (V1).
5. History or family history of inflammatory bowel disease (Crohn's disease or ulcerative colitis) or other conditions characterized by severe intestinal ulcers.
6. History or family history of coeliac disease.
7. Patients with intestinal obstruction or partial intestinal obstruction.
8. Presence of diarrhoea associated with fever and/or blood in the stool.
9. Health conditions requiring continuous or intermittent treatment with facial topical, inhaled or systemic steroids and/or biologic or non-biologic immunosuppressive or immunomodulatory agents (e.g. autoimmune diseases, etc.).
10. Severe kidney impairment (i.e. estimated glomerular filtration rate <30 ml/min).
11. Severe hepatic impairment (i.e. Child-Pugh B or C).
12. Cancer or any cancer-related treatment within 5 years prior to screening (excluding non-melanoma skin-cancer).
13. History of alcohol or drug abuse within a year prior to screening.
14. Facial skin conditions that can interfere with reliable assessment of rosacea throughout the study (e.g. keloids, hypertrophic scarring, recent facial surgery etc.)
15. Any other significant health condition (e.g. cardiovascular, respiratory, renal, hepatic, neurologic, psychiatric, hematologic, oncologic, immune etc.) that in the investigator's judgement may: i) jeopardize the patient's safe participation in the trial or ii) make unlikely the patient's completion of the study or iii) make unlikely the patient's compliance with the study procedures (e.g. highly anticipated need of non-permitted treatments, terminal illness, etc.).
16. History of hypersensitivity to rifaximin, rifamycin-derivatives, any of the rifaximin-EIR excipients, or any UV protection cream component.
17. Treatment with biologic immunomodulatory and/or immunosuppressive drugs (e.g. anti-TNF drugs) within 6 months prior to randomization.
18. Treatment with non-biologic immunomodulatory and/or immunosuppressive drugs (e.g. cyclosporine, methotrexate etc.) within 30 days prior to randomization.
19. Treatment with warfarin within 14 days prior to randomization.
20. Treatment with niacin within 30 days prior to randomization.
21. Topical facial or systemic antibiotics within 30 days before randomization;
22. Treatment with neomycin or other low-absorbable oral antibiotics (such as marketed rifaximin) within 90 days before randomization.
23. Topical facial, inhaled or systemic corticosteroids within 30 days prior to randomization.
24. Topical facial retinoids within 30 days before randomization.
25. Systemic retinoids within 6 months before randomization.
26. Any other topical or systemic treatment for rosacea within 30 days before randomization (including also laser and pulsed light, etc.).
27. Pharmaceutical prebiotics and probiotics (functional food is allowed), within 30 days before randomization.
28. Any experimental treatment within 6 months prior to randomization.
29. Women who are pregnant, breast-feeding or planning a pregnancy during the trial period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline (day 1) in number of rosacea inflammatory lesions (papules, pustules or plaques) at the end of treatment visit (day 30 ± 1) | 30 days
  changes in number of lesions
Percent of participants showing treatment success (IGA score of 0 [clear] or 1 [almost clear]) at the end of treatment visit (day 30 ± 1) | 30 days
  per cent changes in IGA score 0 and 1 patients

SECONDARY OUTCOMES:
Mean change from Baseline (day 1) in number of rosacea inflammatory lesions at the end of treatment visit (day 30 ± 1) as provided by Canfield Image Analysis | 30 days
  changes respect to baseline
Mean change from Baseline (day 1) in number of inflammatory lesions (papules, pustules or plaques) at day 10 ± 1 and day 60 ± 3 | 10 and 60 days
  change respect to baseline
Percent of participants showing treatment success (i.e. IGA score of 0 or 1) at day 10 ± 1 and day 60 ± 3 | 10 and 60 days
  per cent changes in IGA score 0 and 1 patients
Percent of participants with IGA score of 0 (clear) at day 10 ± 1, day 30 ± 1 and day 60 ± 3 | 10, 30 and 60 days
  per cent changes in IGA score 0 patients
Mean change from Baseline (day 1) in the following rosacea additional features at day 10 ± 1, day 30 ± 1 and day 60 ± 3: • burning or stinging • telangiectasia • ocular manifestations • phymatous changes | 10, 30 and 60 days
  change respect to baseline
Mean change from Baseline (day 1) in facial non-transient erythema at day 10 ± 1, day 30 ± 1 and day 60 ± 3 (absent=0, mild=1, moderate=2, severe=3) | 10, 30 and 60 days
  change respect to baseline
Mean change from Baseline (day 1) in number of inflammatory lesions at day 10 ± 1 and day 60 ± 3 as provided by Canfield Image Analysis | 10 and 60 days
  change respect to baseline
Mean change from Baseline (day 1) in facial non-transient erythema score at day 10 ± 1, day 30 ± 1 and day 60 ± 3, based on global fractional area redness as provided by Canfield Image Analysis | 10, 30 and 60 days
  change respect to baseline
Mean change from Baseline in Basic Self-Esteem Scale at day 30 ± 1 and day 60 ± 3 | 30 and 60 days
  change respect to previous evaluation
Mean change from Baseline (day 1) in Dermatology Life Quality Index (10-item DLQI) at day 30 ± 1 and day 60 ± 3 | 30 and 60 days
  change respect to baseline
Mean difference in Treatment Satisfaction Questionnaire between study groups at day 30 ± 1 | 30 days
  differences between treatment arms

OTHER OUTCOMES:
Mean change from Baseline (day 1) in circulating inflammatory marker levels at 10 ± 1, day 30 ± 1 and day 60 ± 3 | 10, 30 and 60 days
  change respect to baseline
Mean change from baseline (day 1) skin texture index at 10 ± 1, day 30 ± 1 and day 60 ± 3 as provided by Canfield Image Analysis | 10, 30 and 60 days
  change respect to baseline

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Ospedali Riuniti di Ancona, Ancona
  - Policlinico di Bari, Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Spedali Civili, Brescia
  - Policlinico Vittorio Emanuele, Catania
  - Ospedale Policlinico San Martino, Genova
  - Ospedale della Misericordia, Grosseto
  - Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Policlinico Universitario A. Gemelli, Roma
  - Azienda Ospedaliera Santa Maria, Terni
  - A.O.U. Città della Salute e della Scienza, Torino